CLINICAL TRIAL: NCT06441760
Title: Efficacy of Teleconsultation to Improve Prehospital Patient Safety for Critically Ill Infants and Children - A Multicenter, Simulation-based Randomized Control Trial
Brief Title: Simulation Trial of Telemedical Support for Paramedics
Acronym: R01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-44972; 1R01HD115574-01 (NIH)
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Emergencies; Cardiopulmonary Arrest; Acute Respiratory Failure; Status Epilepticus
Keywords: Prehospital emergency care; Emergency medical services (EMS); Paramedics; Infant simulator mannequins; Telemedical support; Critically ill infants and children; Pediatric emergencies
MeSH Terms: conditions — Emergencies; Heart Arrest; Status Epilepticus

STUDY DESIGN:
Intervention Model Description: Single blind, parallel arm, multicenter simulation RCT of prehospital teams from 9 Pediatric Emergency Care Applied Research Network (PECARN) and non-PECARN sites
Who Masked: Outcomes Assessor
Masking Description: All participants will be blinded to the simulated transport scenarios.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teleconsultation video arm with PEM physicians (Experimental): Emergency Medical Services (EMS) providers randomized into this arm will receive video teleconsultation with Pediatric Emergency Medicine (PEM) physicians.
  Interventions: Other: Video teleconsultation
- Audio support arm with EM physicians (Active Comparator): EMS providers randomized into this arm will receive audio support by usual care Emergency Medicine (EM) physicians.
  Interventions: Other: Audio support

INTERVENTIONS:
Other: Video teleconsultation — Each team will participate in 4 video-recorded simulated transports in fully equipped ambulances. Each team will provide resuscitative care in 4 simulated high-risk pediatric transports. EMS personnel will provide care in the ambulance while PEM physicians will provide medical direction remotely using video to communicate with EMS personnel via tablet devices.
  Arms: Teleconsultation video arm with PEM physicians
Other: Audio support — Each team will participate in 4 video-recorded simulated transports in fully equipped ambulances. Each team will provide resuscitative care in 4 simulated high-risk pediatric transports. EMS personnel will provide care in the ambulance while EM physicians will provide medical direction remotely using audio to communicate with EMS personnel via tablet devices.
  Arms: Audio support arm with EM physicians

SUMMARY:
In the United States, the current standard of prehospital (i.e. outside of hospitals) emergency care for children with life-threatening illnesses in the community includes remote physician support for paramedics providing life-saving therapy while transporting the child to the hospital. Most prehospital emergency medical services (EMS) agencies use radio-based (audio only) communication between paramedics and physicians to augment this care. However, this communication strategy is inherently limited as the remote physician cannot visualize the patient for accurate assessment and to direct treatment.

The purpose of this pilot randomized controlled trial (RCT) is to evaluate whether use of a 2-way audiovisual connection with a pediatric emergency medicine expert (intervention = "telemedical support") will improve the quality of care provided by paramedics to infant simulator mannequins with life threatening illness (respiratory failure). Paramedics receiving real-time telemedical support by a pediatric expert may provide better care due to decreased cognitive burden, critical action checking, protocol verification, and error correction. Because real pediatric life-threatening illnesses are rare, high stakes events and involve a vulnerable population (children), this RCT will test the effect of the intervention on paramedic performance in simulated cases of pediatric medical emergencies.

The two specific aims for this research are:

* Aim 1: To test the intervention efficacy by determining if there is a measurable difference in the frequency of serious safety events between study groups
* Aim 2: To compare two safety event detection methods, medical record review, and video review

ELIGIBILITY:
Inclusion Criteria:

* Certified Emergency Medical Technicians (EMTs), Advanced EMTs (AEMTs), and Paramedics (EMT-Ps) who provide direct scene response.
* Board-certified Pediatric Emergency Medicine (PEM) and Emergency Medicine (EM) physicians whose practice includes online medical support for EMS are eligible.
* The control arm will include physicians who provide radio/telephone support in usual care at each site. In the intervention arm, experts will be PEM with/without EMS board-certification as they have relevant pediatric training and experience.

Exclusion Criteria:

* EMS personnel providing interfacility transport and/or pediatric specialty transport
* Resident physicians-in-training
* Non-physician providers

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of Serious Safety Events | Post treatment usually 4 hours
  Serious safety events are defined as clinical care actions that reach the patient and have the potential to cause moderate-to-severe harm or death. An investigator developed predefined serious safety event checklist developed for each simulated transport scenario will be used to record serious safety events. Serious safety events will be scored as: present, absent, or not observable.

SECONDARY OUTCOMES:
Composite team score | Post treatment usually 4 hours
  The composite team performance score is calculated from the modified Lammer's simulation checklist tool as the percentage of completed actions that can be observed during the simulation by either video review or in person observation. This checklist tool contains 171 items across 3 simulated transport scenarios that represent critical actions expected for optimal care performance.
Error in medication choice | Post treatment usually 4 hours
  Errors in medication choice are measured by specific items within the modified Lammer's simulation checklist tool. These will be any incorrect type of medication used by a team during simulation, including unanticipated medication choices which raters feel was not indicated or potentially harmful by consensus opinion. This will be reported as the proportion or percentage of items scored as incomplete over all possible items related to medication choice.
Error in weight-based medication dosing | Post treatment usually 4 hours
  These are measured by specific items within modified Lammer's simulation checklist tool. These will be any error in pediatric weight-based dose calculation, including error in volume of administered drug. This will be reported as the proportion or percentage of items scored as incomplete over all possible items related to weight-based medication dosing.
Equipment size error | Post treatment usually 4 hours
  These are measured by specific items within the modified Lammer's simulation checklist tool. These will be any error in size of equipment used during each case. This will be reported as the proportion or percentage of items scored as incomplete over all possible items related to equipment sizing
EMS protocol error | Post treatment usually 4 hours
  These are measured by specific items within the modified Lammer's simulation checklist tool. These will be any error observed omission, error, or deviation in offline and online EMS treatment protocols that could result in patient harm. This will be reported as the proportion or percentage of items scored as incomplete over all possible items related to selection of appropriate EMS protocols.
Equipment Use Error | Post treatment usually 4 hours
  These are measured by specific items within the modified Lammer's simulation checklist tool. These will be any error in equipment usage during each case. This will be reported as the proportion or percentage of items scored as incomplete over all possible items related to equipment use.

CONTACTS AND LOCATIONS:
Overall Officials: Tehnaz Boyle, MD PhD, Principal Investigator — Bosotn Medical Center, Pediatrics Department
Locations (4):
- United States (4):
  - Children's Hospital Colorado, University of Colorado Denver Anschutz Medical Campus, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - BostonMedical Center, Boston, Massachusetts
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No